CLINICAL TRIAL: NCT05159622
Title: Increasing Tap Water Drinking Behaviors Among Young Latino Children-(CentroNia)
Brief Title: Water Up@ At Home: An Intervention to Replace Sugary Drinks With Water
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Uriyoan Colon-Ramos, Associate Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 051719; 5R21DK119749 (NIH)
Record Dates: First submitted 2019-07-17; First posted 2021-12-16 (Actual); Results first posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: nutrition; sugar-sweetened beverages; water security; diet; infants; toddlers
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Effect Evaluation: Using a pre- and post-evaluation design, the investigators will evaluate the effects of randomized controlled trial by comparing self-reported SSB intake (servings/day) among participants in the intervention vs. control groups. Data collection points are: baseline, follow-up (12-weeks after the start of the intervention), and a second follow-up (12 months after the start of the intervention) to explore the sustainability of behaviors and potential effect on anthropometric measures. The entire survey (lasting about 40 minutes) will be administered at home.
  Primary Outcome (SSB intake) During the three data collection periods, the investigators will use the Beverage Intake Questionnaire a quantitative food frequency questionnaire that assesses habitual beverage consumption of 15 beverage categories in the past month.
Who Masked: Outcomes Assessor
Masking Description: Data collector will not know if the participant received the intervention or control curriculum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Description of behavioral intervention Water Up! at Home: The intervention is theory-based and was designed to be sensitive to the context, perceptions and needs of this high risk population. It was collaboratively developed with key stakeholders in the predominantly Latino immigrant community. The curriculum consists of 12 infographics and lessons (bilingual Spanish/English) designed to increase knowledge of drinking water health benefits, safety/cleanliness, cost/convenience, prior experience. The 12-week intervention will be delivered in participants' home by the home visitor. Participants will receive a water filter for use in their home in addition to educational information about water and sugary beverages. Throughout the lessons, they will be asked to complete various activities such as taking pictures and engaging in discussions about their water drinking habits.
  Interventions: Behavioral: Water Up! at Home
- Control (No Intervention): Participants will receive the standard educational curriculum from the home visiting program (and also a water filter as a token of appreciation).

INTERVENTIONS:
Behavioral: Water Up! at Home — 1: Addressing physical barriers to replace SSB with water at home: Participants will receive a personal, reusable bottle of water, a National Sanitation Foundation-certified water filter pitcher and one additional filter cartridge 2: Addressing sociocultural barriers to change individual perceptions: The curriculum has 6 topics delivered in 12 sessions: a) water for your health (diabetes/obesity among Latinos); b) health benefits of water vs. SSB, c) sugar content of SSB, d) safety & affordability of filtered tap water vs. bottled beverages, e) access and promotion of SSB vs. water in your community, f) tips for improving water taste, perceived susceptibility, severity, costs and benefits. 3: Addressing sociocultural barriers to increase skills: During each session, participants will be asked to perform hands-on learning activities (e.g., measure sugar content in SSB, take pictures of themselves explaining to their family members the key messages of various lessons).
  Arms: Intervention

SUMMARY:
This study will test the preliminary effects of an intervention to reduce sugary drinks among low-income parents (n=38)(primary caregivers) and their young children (6 months-3 year olds) compared to a control group (n=38). The main outcome is behavioral: sugary drink consumption (self-reported servings/day) among parents and among their children (parent-reported servings/day). These outcomes are measured at baseline and immediately after the 12-week intervention. An exploratory aim will test if the intervention has a sustained behavioral effect and an effect on body mass index and waist circumference of the parents 12 months after baseline.

Our mixed methods multi-phase approach includes a quantitative component (randomized controlled trial - Aim 1) and a qualitative component (in-depth interviews and focus groups- Aim 2) to test the effects of a behavioral intervention to replace sugary drinks with water at home.

DETAILED DESCRIPTION:
Consumption of sugar-sweetened beverages (SSB) is a risk factor for obesity, diabetes, and other chronic diseases. Consumption of SSB begins at an early age and may have cumulative detrimental consequences to health later in life. There is an urgent need to facilitate reduction of SSB consumption among young children before this behavior becomes part of an unhealthy lifestyle. The public health recommendation to drink water instead of SSB does not consider the multiple barriers that underserved communities face when choosing a beverage in an environment with limited access to clean, palatable drinking water, and saturated with SSB promotion. Using a community participatory approach, the investigators developed an intervention, Water Up! at Home, which draws on theory and community experience to position parents as social models for their young children. The objective of the current proposal is to test the preliminary effects of this intervention to replace SSB with filtered tap water among low-income parents and their children (6 months-3 year olds). The working hypothesis is that by addressing sociocultural (via curriculum) and physical (via water filter) barriers, parents can reduce their own and their children's SSB consumption. The investigators will use a multiphase sequential mixed-methods design to integrate qualitative and quantitative findings. Aim 1) Partnering with an existing home visiting program of Early Head Start (EHS), the EHS staff will deliver the intervention to replace SSB with filtered tap water at home and test its effects using a randomized control trial. H1) Parents randomly assigned to the Water Up! at Home program (n=38) will see a net reduction of 0.5 servings/day of SSB compared with the control group at the end of the intervention (12 weeks). H2) Findings will show a similar reduction in SSB consumption among young children. Exploratory aim: 12 months after baseline, the investigators will explore changes on body mass index and waist circumference of parents. To assess the quality of program implementation, the investigators will use a summative process evaluation. Aim 2) To assess the psychosocial mediators of intervention effects and to understand why the program was or was not successful, the investigators will conduct 30 in-depth interviews with parents, segmented by whether they responded positively/negatively to the intervention. The investigators will also conduct two focus groups with Early Head Start staff (n=10) to describe the aspects of the intervention design, context, implementation and delivery that may affect program impact, its sustainability and practicability. The study addresses a novel paradigm that posits water security at home as a determinant of SSB consumption among low-income parents and their children.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 year old) primary caregivers (biological parents, legal guardians) with at least 1 child enrolled in the CentroNia home-visiting program.
* No intention of moving from the neighborhood or moving out of the program for the next year

Exclusion Criteria:

* Caregivers with children younger than 6 months old at time of recruitment.
* Caregivers who have access or be using a water filtration system including pitchers with filters or an installed filtering device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santillan-Vazquez C, Hernandez L, Reese AC, Burgos-Gil R, Cleary SD, Rivera IM, Gittelsohn J, Edberg MC, Monge-Rojas R, Colon-Ramos U. How providing a low-cost water filter pitcher led Latino parents to reduce sugar-sweetened beverages and increase their water intake: explanatory qualitative results from the Water Up!@Home intervention trial. Public Health Nutr. 2022 Nov;25(11):3195-3203. doi: 10.1017/S1368980022001744. Epub 2022 Aug 19. PMID 35983682
- [Derived] Reese AC, Burgos-Gil R, Cleary SD, Lora K, Rivera I, Gittelsohn J, Seper S, Monge-Rojas R, Colon-Ramos U. Use of a Water Filter at Home Reduces Sugary Drink Consumption among Parents and Infants/Toddlers in a Predominantly Hispanic Community: Results from the Water Up!@ Home Intervention Trial. J Acad Nutr Diet. 2023 Jan;123(1):41-51. doi: 10.1016/j.jand.2022.06.006. Epub 2022 Jun 15. PMID 35714910

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult parents (>18 yrs of age) of children aged 6 months to 3 yrs old who were enrolled in the home-visiting program of three Early Head Start centers in the Washington District of Columbia (DC) metropolitan area were eligible to participate in the study. After screening for eligibility criteria with the assistance of Early Head Start home visitors, a bilingual (Spanish/English) and trained data collector called eligible families to invite them to participate in the study and consent them.
Pre-assignment Details: There were no significant events after participant enrollment. In terms of recruitment, 101 parents were originally recruited and completed a baseline survey but prior to assignment to groups, nine of those parents were deemed ineligible for the following reasons: the children of 6 parents aged out of the home visiting program; the children of 3 parents were younger than 6 months of age at time of recruitment and therefore not enrolled.
Groups:
- Intervention Water Up!@Home: Participants received a BPA-free infusion water bottle, a child-size pitcher to be used for serving water, and a National Sanitation Foundation-certified 11-cup low-cost water filter pitcher and one additional filter cartridge.
  A 12-session curriculum delivered weekly by home visitors at home of participants included hands-on activities that emphasized observational learning, parent-child modeling of behaviors in beverage choice, and modeling behaviors to offer filtered tap water instead of juice or sugary drinks, and weekly goal setting to replace or dilute selected sugary drinks for themselves and their child.
- Comparison: During the same 12 weeks, comparison participants received the standard weekly educational curriculum from the home visiting program and the same low-cost water filter pitcher was provided as a token of appreciation).
Period: Overall Study
Arm/Group | Intervention Water Up!@Home | Comparison
Started | 45 | 47
Completed | 41 | 42
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Intervention Water UP!@Home: 12 week intervention and low-cost water filter pitcher
- Comparison: Standard educational curriculum from the home visiting program and also a water filter pitcher as a token of appreciation.
- Total: Total of all reporting groups
Arm/Group | Intervention Water UP!@Home | Comparison | Total
Number analyzed (Participants) | 45 | 47 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (6.8) | 32.3 (7) | 32.03 (7.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 45 | 87
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 47 | 92
Language of preference: Spanish [Count of Participants; unit: Participants] | 37 | 40 | 77
Parent-reported sex of their child: female [Count of Participants; unit: Participants] | 26 | 23 | 49
Country of birth [Count of Participants; unit: Participants]
  United States | 14 | 6 | 20
  Guatemala | 14 | 18 | 32
  El Salvador | 4 | 8 | 12
  Mexico | 1 | 3 | 4
  Ethiopia | 8 | 4 | 12
  Other | 3 | 6 | 9
  Nicaragua | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Sugary Drink Consumption for Parents
Description: Amount of sugary drinks consumed (ounces) per day. Sugar-sweetened beverages was a composite variable created from the sum of sweetened fruit drink, soda, flavored milk, sweetened coffee/tea, and sports or energy drinks.
Time Frame: Baseline, post-treatment starting 12 weeks after start of intervention, and at most 16 weeks after start of intervention
Population: Parents (adults> 18 yrs of age) who completed the intervention.
Measure: Median (Full Range); unit: oz/day
Groups:
- Intervention Water Up!@Home: The intervention was informed by formative research, and combined elements of the Social Cognitive Theory and the Health Belief Model to address both physical (perceptions of tap water quality and safety) and sociocultural barriers to replacing sugary drinks and excess juice consumption with water, primarily from tap.
  Participants received a BPA-free infusion water bottle, a child-size pitcher to be used for serving water, and a National Sanitation Foundation-certified 11-cup low-cost water filter pitcher and one additional filter cartridge.
  A 12-session curriculum delivered weekly by home visitors at home of participants included hands-on activities that emphasized observational learning, parent-child modeling of behaviors in beverage choice, and modeling behaviors to offer filtered tap water instead of juice or sugary drinks, and weekly goal setting to replace or dilute selected sugary drinks for themselves and their child. Home visits conducted in 10-35 min of the 90 min Early Head Start standard home visit.
Arm/Group | Intervention Water Up!@Home | Comparison
Number analyzed (Participants) | 45 | 47
oz/day
  Baseline oz/day median | 12 [0 to 96] | 14.29 [0 to 88]
  Endline oz/day median | 4.57 [0 to 53.5] | 8.57 [0 to 48.28]
Statistical Analysis 1: Comparison: Intervention Water Up!@Home vs Comparison; Test type: Equivalence — A net effect of 6 fluid oz/day (SD=1) was hypothesized among adult parents, assuming two sided alpha=0.05, power = 80%, and a minimum sample size of 60 adults; p = 0.15, t-test, 2 sided — The a priori threshold for statistical significance is <0.05. P-value of the interaction between treatment group and change in beverage consumption (fl oz/day); Median Difference (Final Values) = 3.2

2. Primary Outcome: Change in Water Consumption for Parents
Description: Change in the amount of water consumed in oz/day from baseline
Time Frame: baseline, post-treatment starting 12 weeks after start of intervention and at most 16 weeks after start of intervention
Population: Parent (adults > 18 yrs old) who completed baseline data collection, endline data collection.
Measure: Median (Full Range); unit: oz/day
Arm/Group | Intervention Water Up!@Home | Comparison
Number analyzed (Participants) | 45 | 47
oz/day
  Median fluid oz/day at baseline | 27 [6 to 87] | 48 [.86 to 60]
  Median fluid oz/day at endline: number analyzed (Participants) | 41 | 42
  Median fluid oz/day at endline | 38.14 [14.9 to 85.7] | 36.43 [18 to 108]
Statistical Analysis 1: Comparison: Intervention Water Up!@Home vs Comparison; Test type: Equivalence — This was an exploratory outcome; p = 0.98, t-test, 2 sided; Median Difference (Final Values) = 0.07

3. Secondary Outcome: Parent-reported Water Consumption of Their Infant/Toddler
Description: Parents were asked to report on the water consumption of their infant/toddler at baseline and endline.
Time Frame: Up to 16 weeks from baseline
Population: Parents, who report on their infants/toddlers' beverage consumption
Measure: Median (Full Range); unit: oz/day
Groups:
- Intervention Water Up!@Home: The intervention was informed by formative research, and combined elements of the Social Cognitive Theory and the Health Belief Model to address both physical (perceptions of tap water quality and safety) and sociocultural barriers to replacing sugary drinks and excess juice consumption with water, primarily from tap.
  Participants received a BPA-free infusion water bottle, a child-size pitcher to be used for serving water, and a National Sanitation Foundation-certified11-cup low-cost water filter pitcher and one additional filter cartridge.
  A 12-session curriculum delivered weekly by home visitors at home of participants included hands-on activities that emphasized observational learning, parent-child modeling of behaviors in beverage choice, and modeling behaviors to offer filtered tap water instead of juice or sugary drinks, and weekly goal setting to replace or dilute selected sugary drinks for themselves and their child. Home visits conducted in 10-35 min of the 90 min Early Head Start standard home visit.
Arm/Group | Intervention Water Up!@Home | Comparison
Number analyzed (Participants) | 45 | 47
oz/day
  Median water intake at baseline (oz/day) infants/toddlers (parent reported) | 6 [0 to 36] | 6 [0 to 19]
  Median water intake at endline (oz/day) infants/toddlers (parent reported): number analyzed (Participants) | 41 | 42
  Median water intake at endline (oz/day) infants/toddlers (parent reported) | 8 [1.43 to 37.5] | 7.36 [1.43 to 30]
Statistical Analysis 1: Comparison: Intervention Water Up!@Home vs Comparison; Test type: Equivalence — This was an exploratory outcome and therefore statistical power was not based on a hypothesis of this outcome; p = 0.36, t-test, 2 sided; Median Difference (Final Values) = 0.64

4. Secondary Outcome: Parent-reported Sugary Drink Consumption of Their Infant/Toddler
Description: Parents were asked to report on their infant/toddlers' beverage consumption at baseline and endline.
Time Frame: Baseline and up to 16 weeks after baseline
Population: Parents' report of their infant/toddler beverage consumption
Measure: Median (Full Range); unit: oz/day
Groups:
- Intervention Water Up!@Home: The intervention was informed by formative research, and combined elements of the Social Cognitive Theory and the Health Belief Model to address both physical (perceptions of tap water quality and safety) and sociocultural barriers to replacing sugary drinks and excess juice consumption with water, primarily from tap.
  Participants received a BPA-free infusion water bottle, a child-size pitcher to be used for serving water, and a National Sanitation Foundation-certified PUR 11-cup low-cost water filter pitcher and one additional filter cartridge.
  A 12-session curriculum delivered weekly by home visitors at home of participants included hands-on activities that emphasized observational learning, parent-child modeling of behaviors in beverage choice, and modeling behaviors to offer filtered tap water instead of juice or sugary drinks, and weekly goal setting to replace or dilute selected sugary drinks for themselves and their child. Home visits conducted in 10-35 min of the 90 min Early Head Start standard home visit.
Arm/Group | Intervention Water Up!@Home | Comparison
Number analyzed (Participants) | 45 | 47
oz/day
  Baseline (oz/day) Parent-reported sugary drink consumption for infants/toddlers | 0 [0 to 28.5] | 0.29 [0 to 25.72]
  Endline- oz/day parent-report on sugary drink consumption of their infants/toddlers: number analyzed (Participants) | 41 | 42
  Endline- oz/day parent-report on sugary drink consumption of their infants/toddlers | 0 [0 to 22.5] | 0.14 [0 to 20]
Statistical Analysis 1: Comparison: Intervention Water Up!@Home vs Comparison; Test type: Equivalence — Exploratory outcome as for infants/toddlers based on parent-report; p = 0.92, t-test, 2 sided; Median Difference (Final Values) = 0.14

5. Secondary Outcome: Parent-reported 100% Fruit Juice Consumption for Their Infant/Toddler
Description: Parent-reported 100% fruit juice consumption for their infant/toddler at baseline and at endline
Time Frame: Baseline and up to 16 weeks after baseline
Population: Parents who reported on their infant and toddler consumption of beverages
Measure: Median (Full Range); unit: oz/day
Arm/Group | Intervention Water Up!@Home | Comparison
Number analyzed (Participants) | 45 | 47
oz/day
  Baseline | 0.71 [0 to 15] | 1.79 [0 to 15]
  Endline: number analyzed (Participants) | 41 | 42
  Endline | 0.71 [0 to 7.50] | 1.79 [0 to 10]
Statistical Analysis 1: Comparison: Intervention Water Up!@Home vs Comparison; Test type: Equivalence — Exploratory outcome; p = 0.03, t-test, 2 sided; Median Difference (Final Values) = 0.95

6. Secondary Outcome: Parent 100% Fruit Juice Consumption
Description: Amount of 100% fruit juice consumed (ounces) per day.
Time Frame: From baseline up to 16 weeks
Population: Parents who completed the baseline and endline surveys.
Measure: Median (Full Range); unit: oz/day
Arm/Group | Intervention Water Up!@Home | Comparison
Number analyzed (Participants) | 45 | 47
oz/day
  Baseline | 2.86 [0 to 24] | 2.86 [0 to 36]
  Endline: number analyzed (Participants) | 41 | 42
  Endline | 0 [0 to 12] | 2.86 [0 to 16]

7. Other Pre Specified Outcome: Body Mass Index for Parents
Description: These measures were only collected at baseline, due to challenges from the onset of the COVID-19 pandemic. At baseline, body weight and body height were measured twice from parents who were barefoot and wearing light clothing, standing on the center of the scale and in a vertical position, using a scale with precision of 100g, and a stadiometer (for weight). Body mass index was calculated from kg/m^2.
Time Frame: Baseline
Population: Participants were adults (>18 yrs old) from cohort 1 (pre-pandemic) randomized to either intervention or comparison group.
Measure: Mean (Standard Deviation); unit: kg/m(2)
Groups:
- Intervention Water Up!@Home; Comparison: Baseline data on this indicator was collected only at baseline due to COVID-19 pandemic onset. Therefore, here we do not describe the intervention.
Arm/Group | Intervention Water Up!@Home | Comparison
Number analyzed (Participants) | 31 | 33
kg/m(2) | 29.4 (6.1) | 29.6 (6.5)

8. Other Pre Specified Outcome: Waist Circumference for Parents
Description: This was only collected at baseline from some participants due to the onset of COVID-19. At baseline Measured from parents in a standing position, at midpoint between the lower border of the last rib and the upper border of the iliac crest on the horizontal place, using an inextensible Gulick measuring tape graduated in cm. Data collectors took 3 waist circumference measurements (the average was used for analyses).
Time Frame: Baseline
Population: Adults (>18 yrs old) who completed baseline data collection.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intervention Water Up!@Home | Comparison
Number analyzed (Participants) | 31 | 33
cm | 88.1 (12.3) | 89.8 (12.5)

9. Other Pre Specified Outcome: Hip Circumference for Parents
Description: Measured from parents in a standing position, at midpoint on the widest part of the hips, horizontal place, using an inextensible Gulick measuring tape graduated in cm. Data collectors took 3 hip circumference measurements (the average was used for analyses).
Time Frame: Baseline
Population: Adult parents (>18 yrs old) who completed baseline data collection
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Intervention Water Up!@Home: Only collected at baseline due to COVID-29
- Comparison: Only collected at baseline due to COVID-19
Arm/Group | Intervention Water Up!@Home | Comparison
Number analyzed (Participants) | 31 | 33
cm | 108.2 (11.4) | 106.2 (13.7)

ADVERSE EVENTS:
Time Frame: Serious and other adverse event data and all-cause mortality were not collected/monitored systematically. The research team met weekly or daily during data collection to review data quality, discuss and resolve any issues with data collection or reporting problems, and discuss any sensitivity or participant reactions to data collected and data collection procedures. Participants were all parents (adults > 18 yrs of age). Adverse events were also not monitored for children.
Description: Serious and other [non-serious] adverse events were not collected or assessed as part of the study. The definition for adverse event/serious adverse event did not differ from clinicaltrials.gov definition.
Groups:
- Intervention Water Up!@Home; Comparison: Serious and other [non-serious] adverse events were not collected or assessed as part of the study).
Arm/Group | Intervention Water Up!@Home | Comparison
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT05159622/Prot_SAP_000.pdf